CLINICAL TRIAL: NCT06761872
Title: Predisposing Factors and Prevalence of Pericardial Diseases Among ESRD Patients Who Are Admitted in Critical Care Medicine Unit in Assuit University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Elsayed, Resident Physician, Assiut University
Other Study IDs: Pericardial disease in ESRD pt
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Pericardial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objectives of this observational study are:

1. Provide reliable data on the prevalence of pericardial diseases, pericardial effusion, constrictive pericarditis and its predisposing factors among ESRD patients, undergoing long-term dialysis.
2. Detect the predisposing factors that could contribute to pericardial effusion amount and severity.

Participants (or their designated contact persons) will be contacted over the phone for either a telephone interview or a follow-up visit in the outpatient clinics, whatever feasible and possible.

DETAILED DESCRIPTION:
* Inclusion Criteria: Patients with ESRD with a GFR <10 cc/min admitted to the internal medicine department nephrology unit or undergoing regular hemodialysis.
* Exclusion Criteria: Patients presented with non-uremic pericarditis such as intra-thoracic malignancy, injury (thoracic, oesophageal, and iatrogenic trauma), pulmonary TB, autoimmune diseases, history suggestive of recent viral infection, myxedema, and severe HF.
* Study tools:

  1. Demographic data (age, sex, and comorbidities).
  2. Clinical data including (The etiology of ESRD). (History of stitching anterior chest pain worse on inspiration, audible friction rub, and raised JVP).

     (Muffled heart sounds, ascites, and lower limb edema).
  3. ECG for signs of pericarditis, such as concave ST segment elevation in all leads, and signs of tamponade, such as low-voltage complexes with electrical alternates.
  4. Doppler echocardiography by Phillips HD 11: for detection of amount and severity of pericardial effusion. The severity was defined as Small (10 < mm echo-free space behind the left ventricle). Moderate (10-20 mm, echo-free space behind the left ventricle and in front of the right ventricle in less than 1 cm).

     Large (>20 mm which was the mentioned finding in addition to a right-sided atrial collapse).
  5. Echocardiography in constrictive pericarditis shows the presence of small left ventricular dimensions with preserved systolic function, impaired diastolic function, dilated atria, abrupt termination of diastolic filling, interventricular septal bounce expiratory diastolic flow reversal in hepatic veins and tissue doppler of the medial mitral annulus is more than lateral.
  6. Serum calcium and phosphorus concentrations and creatinine levels in both serum and urine were elevated. Serum lipid profile, serum albumin, hormone tests such as thyroid and parathyroid along with complete blood count.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD with a GFR <10 cc/min are admitted to the internal medicine department nephrology unit or undergoing regular hemodialysis.

Exclusion Criteria:

* Patients presented with non-uremic pericarditis such as intra-thoracic malignancy, injury (thoracic, oesophageal, and iatrogenic trauma), pulmonary TB, autoimmune diseases, history suggestive of recent viral infection, myxedema, and severe HF.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ESRD with a GFR <10 cc/min are admitted to the internal medicine department nephrology unit or undergoing regular hemodialysis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Detection of variable pericardial diseases in patients with ESRD. | 1 year
  variable pericardial diseases in patients with ESRD.

SECONDARY OUTCOMES:
Detection of predisposing factors of pericardial effusion. | 1 year
  predisposing factors of pericardial effusion.

IPD SHARING:
Plan to Share IPD: No